CLINICAL TRIAL: NCT06245200
Title: UNIPDES- An Internet-Based Transdiagnostic Intervention for College Students' Psychological Symptoms: Evaluation of Its Development, Usability and Effectiveness Study Protocol
Brief Title: UNIPDES- An Internet-Based Transdiagnostic Intervention for College Students' Psychological Symptoms
Acronym: UNIPDES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anadolu University (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-80558721-050.99-2300154653; 123K895 (Other Grant/Funding Number: THE SCIENTIFIC AND TECHNOLOGICAL RESEARCH COUNCIL OF TÜRKİYE)
Record Dates: First submitted 2024-01-21; First posted 2024-02-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue
Keywords: cognitive behavioral therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Internet Based Intervention (Experimental): Participants in this group will use the UNIPDES intervention with guidance support.
  Interventions: Other: UNIPDES - Internet Based Intervention - GUIDED
- Unguided Internet Based Intervention (Experimental): Participants in this group will use the UNIPDES intervention without guidance
  Interventions: Other: UNIPDES - Internet Based Intervention - UNGUIDED
- Waitlist (No Intervention): Participants in this group will not receive any intervention. However, if they wish, they will be able to access the UNIPDES unguided version when the trial ends.

INTERVENTIONS:
Other: UNIPDES - Internet Based Intervention - GUIDED — The experimental group participants will receive the internet-based intervention consisting of six weeks. This intervention has cognitive, emotional and behavioral components. Users will be able to use content created with video, audio, animation and interactive forms on their electronic devices (PC; tabs or smartphones). Participants in this arm will receive weekly feedback from counselors through the web software used.
  Arms: Guided Internet Based Intervention
Other: UNIPDES - Internet Based Intervention - UNGUIDED — The experimental group participants will receive the internet-based intervention consisting of six weeks. This intervention has cognitive, emotional and behavioral components. Users will be able to use content created with video, audio, animation and interactive forms on their electronic devices (PC; tabs or smartphones).
  Arms: Unguided Internet Based Intervention

SUMMARY:
This study is a randomised clinical trial. This study evaluates the effect of an internet-based intervention developed based on a transdiagnostic cognitive behavioural approach on psychological symptoms of university students. There are internet-based guided intervention, internet-based unguided intervention and control group in the study.

Experimental group participants (guided and unguided) will use the UNIPDES programme developed within the scope of the project. Participants in the guided internet-based experimental group will additionally receive weekly feedback from the guide .

DETAILED DESCRIPTION:
This study is a randomised clinical trial. This study evaluates the effect of an internet-based intervention developed based on a transdiagnostic cognitive behavioural approach on psychological symptoms of university students. There are internet-based guided intervention, internet-based unguided intervention and control group in the study.

Experimental group participants (guided and unguided) will use the UNIPDES programme developed within the scope of the project. Participants in the guided internet-based experimental group will additionally receive weekly feedback from the guide .

There is a six-week intervention protocol within the programme. This intervention programme includes structured, emotional, cognitive and behavioural interventions independent of the diagnosis.

Users will complete each module in 30-40 minutes. The programme is structured in a hierarchical order. Each session is a preliminary to the session that follows it.

The data will be compared with suitable statistical techniques.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study;
* having a valid e-mail address;
* having internet access (computer or mobile device);
* being over the age of 18;

Exclusion Criteria

* ongoing psychological support/psychotherapy during the research period;
* scoring more than 15 on the Patient Health Questionnaire 9 (PHQ 9) and more than 14 on the Generalized Anxiety Disorder-7 (GAD-7) scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) Turkish Form | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  For asses depression symptoms level. PHQ-9 consists of 9 items structured on a four-point Likert scale (0-3) to measure the level of depressed mood. The lowest score is 0 and the highest score is 27. A high score indicates a high level of depression. It is a self-report tool and participants evaluate themselves.
Generalized Anxiety Disorder-7 (GAD-7) Turkish Form | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  It will use for anxiety symptoms level. The GAD-7 consists of 7 items structured in a four-point Likert scale to measure anxiety level. The lowest score is 0 and the highest score is 21. A high score indicates a high level of anxiety. It is a self-report tool and participants evaluate themselves.
The Brief Adjustment Scale-6 (BASE-6) Turkish Form | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  individual's general psychological distress and adjustment.BASE-6 consists of 6 items structured on a seven-point Likert scale (1-7) to measure the participants' level of adjustment. The lowest score is 7 and the highest score is 42. A high score indicates a high level of negative adjustment and high distress. It is a self-report tool and participants evaluate themselves.

SECONDARY OUTCOMES:
System Usability Scale (SUS-10) Turkish Form: SUS-10 | post-test (6 weeks later from pre-test)
  is a tool aiming to assess the impact of program usability on treatment outcomes. SUS-10 was developed to assess the usability of a system. It consists of 10 items. The items are on a 5-point Likert scale (0-4). The lowest score is 0 and the highest score is 40. A high score indicates high usability. Raw scores are multiplied by 2.5 when calculating. A score above 70 is considered as sufficient usability.

OTHER OUTCOMES:
Attitudes Toward Internet-Based Interventions Scale (ETAM) Turkish Form | Pre-test
  ETAM will use people's opinions/attitudes about internet-based interventions. It consists of 16 items. It is defined as a five-point Likert scale. A high score indicates a positive attitude towards internet-based interventions.
Demographic Information Form | Pre-test
  gather information about the demographics of the participants, including their age, gender, and history of psychiatric treatment/help.
Module Evaluation | during the experiment
  At the end of each module, users will be asked a single question to evaluate the module. With this measurement, it will be assessed how functional the participants find the module. It is scored between 0-10, with a high score indicating that the module is considered functional.
User Experience on Program Effectiveness | post-test (6 weeks later from pre-test)
  Refers to qualitative interviews to be conducted. Interviews will be evaluated by content analysis.

IPD SHARING:
Plan to Share IPD: Yes
Informed consent and study protocol will be shared in the academic journal planned to be published. The data will be forwarded to researchers working in this field upon request from the researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Before the experiment
Access Criteria: open access journal for everyone and request from PI

REFERENCES:
- [Derived] Ozer O, Oztemur G, Altinoz AE, Koksal B, Dogan U, Batmaz S, Gur R, Altinok A. UNIPDES - An internet-based transdiagnostic intervention for college students' psychological symptoms: Evaluation of its development, usability and effectiveness: Study protocol. Contemp Clin Trials Commun. 2025 Feb 6;44:101443. doi: 10.1016/j.conctc.2025.101443. eCollection 2025 Apr. PMID 40191049